CLINICAL TRIAL: NCT03217071
Title: PembroX: Enhancing the Immunogenicity of Non-Small Cell Lung Cancer With Pembrolizumab +/- Stereotactic Radiotherapy Delivered in the Preoperative Window, A Randomized Phase II Study With Correlative Biomarkers
Brief Title: Pembrolizumab With and Without Radiotherapy for Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sue Yom (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Sue Yom, Associate Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 166520; NCI-2017-01727 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2017-07-10; First posted 2017-07-13 (Actual); Results first posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-09

CONDITIONS: Non Small Cell Lung Cancer
Keywords: non small cell lung cancer, resectable
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; Radiosurgery; Surgical Procedures, Operative; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pembrolizumab + Surgery (Experimental): Patients will receive 200mg pembrolizumab on Day 1 of each 3 week cycle, for 2 cycles, prior to surgery. Pembrolizumab will be administered via IV infusion for 30 minutes. Surgery will occur no later than 6 weeks following the last dose of pembrolizumab.
  Interventions: Drug: Pembrolizumab; Procedure: Surgery (Non-interventional, standard of care)
- Pembrolizumab + Radiation + Surgery (Experimental): Patients will receive 200mg pembrolizumab on Day 1 of each 3 week cycle, for 2 cycles. Pembrolizumab will be administered via IV infusion for 30 minutes.Within the week (7 days +/- 3 days) following administration of the second cycle, a single 12 Gy dose of stereotactic radiation therapy (SRT) will be delivered to 50% of the primary tumor only. Definitive surgical resection will occur no later than 6 weeks following the last dose of pembrolizumab.
  Interventions: Drug: Pembrolizumab; Radiation: stereotactic radiation therapy (SRT); Procedure: Surgery (Non-interventional, standard of care)

INTERVENTIONS:
Drug: Pembrolizumab — All study participants will receive pembrolizumab every 3 weeks, for 2 cycles.
  Other Names: Keytruda
Radiation: stereotactic radiation therapy (SRT) — Patients in Cohort 2 of the Safety run-in and patients in the expansion cohort who are randomized to the 'pembrolizumab +radiation arm' will receive one dose of SRT within 1 week (+/- 3 days) following the second administration of pembrolizumab.
  Arms: Pembrolizumab + Radiation + Surgery
Procedure: Surgery (Non-interventional, standard of care) — Standard of care surgery to remove cancer

SUMMARY:
This is a randomized single-institution, phase II, open-label clinical trial of neoadjuvant pembrolizumab with or without low-dose stereotactic radiation therapy (SRT) in stage I-IIIA non-small lung cancer (NSCLC) patients who are planned to undergo surgical resection of their lung cancer.

DETAILED DESCRIPTION:
Two consecutive run-in cohorts will administer pembrolizumab or pembrolizumab with SRT of 12 Gy to the lateral aspect of the primary tumor. Patients will receive pembrolizumab for 2 cycles prior to surgery or SRT and surgery. Surgical resection of all involved areas of tumor will occur within 6 weeks of the last administration of pembrolizumab. It should be noted that surgery is expected to occur within a much shorter window and 6 weeks would represent the greatest allowable amount of delay.

If during the run-in, only the pembrolizumab-alone cohort meets pre-specified safety parameters, subsequently enrolled patients will enter a larger expansion cohort, with treatment given according to that cohort only. If during the run-in both cohorts meet pre-specified safety parameters, subsequently enrolled patients will enter the expansion cohort and be randomized between preoperative pembrolizumab versus pembrolizumab with SRT of 12 Gy.

ELIGIBILITY:
Diagnosis/Condition for Entry into the Trial

1. Histologically or cytologically confirmed non-small cell lung cancer, performed on a biopsy that occurred within the last 60 days.
2. Positron Emission Tomography (PET)-CT within the last 30 days showing radiographic stage I to IIIa lung cancer (mediastinal staging biopsy is allowed but not required).
3. Documentation that the patient is a candidate for surgical resection of their lung cancer by an American Board of Thoracic Surgery-certified surgeon.
4. Measurable disease as defined by RECIST v1.1.
5. Adequate tissue specimens for correlative biomarker analysis. The patient should be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day 1. Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen only upon agreement from the Principal Investigator.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
7. Resolution of all acute toxic effects of prior chemotherapy, radiotherapy or surgical procedures to NCI CTCAE Version 4.0 grade 1.

Inclusion Criteria:

1. Be willing and able to provide written informed consent/assent for the trial.
2. Be at least 18 years of age on day of signing informed consent.
3. Demonstrate adequate organ function as defined below. All screening labs should be performed within 10 days of treatment initiation.

   System Laboratory Value Hematological Absolute neutrophil count (ANC) greater than or equal to 1,500 /microliter (mcL) Platelets greater than or equal to 100,000 / mcL Hemoglobin greater than or equal to 9 g/dL or ≥5.6 mmol/L without transfusion or erythropoietin (EPO) dependency (within 7 days of assessment)

   Renal Serum creatinine OR Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) less than or equal to 1.5 X upper limit of normal (ULN) OR

   Greater than or equal to 60 mL/min for subject with creatinine levels greater than 1.5 X institutional ULN Hepatic Serum total bilirubin Less than or equal to 1.5 X ULN aspartate aminotransferase (AST)/serum glutamic-oxaloacetic transaminase (SGOT), alanine aminotransferase (ALT)/serum glutamic-pyruvic transaminase (SGPT) Less than or equal to 2.5 X ULN

   Coagulation International Normalized Ratio (INR) or Prothrombin Time (PT)

   Activated Partial Thromboplastin Time (aPTT) Less than or equal to 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants Less than or equal to 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants

   Creatinine clearance should be calculated per institutional standard.
4. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
5. Female subjects of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of study medication.

   Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
6. Male subjects of childbearing potential must agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Exclusion Criteria:

1. Is ineligible for an operation based on medical or oncologic contraindications to surgery.
2. Has history of non-infectious pneumonitis/interstitial lung disease that required steroids, or has current pneumonitis/interstitial lung disease.
3. Has evidence of interstitial lung disease.
4. Has an active second malignancy, i.e. patient known to have potentially fatal cancer present for which he/she may be (but not necessarily) currently receiving treatment. Patients with a history of malignancy that has been completely treated, with no evidence of that cancer currently, are permitted to enroll in the trial if curative therapy has been completed, such as basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
5. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
6. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
7. Has a known history of active Bacillus Tuberculosis (TB)
8. Hypersensitivity to pembrolizumab or any of its excipients.
9. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., Less than or equal to Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
10. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., less than or equal to Grade 1 or at baseline) from adverse events due to a previously administered agent.

    * Note: Subjects with less than or equal to Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
    * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
11. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
12. Has an active infection requiring systemic therapy.
13. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
14. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
15. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
16. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
17. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
18. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (HCV) (e.g., HCV RNA [qualitative] is detected).
19. Has received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of the study drug. Administration of killed vaccines is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-10-04 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sue Yom, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pembrolizumab + Surgery | Pembrolizumab + Radiation + Surgery
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab + Surgery | Pembrolizumab + Radiation + Surgery | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Customized [Count of Participants; unit: Participants]
  40-49 years old | 0 | 1 | 1
  50-59 years old | 2 | 1 | 3
  60-69 years old | 3 | 2 | 5
  70-79 years old | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 2 | 4 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 4 | 6 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 1 | 1
  White | 4 | 4 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in the Mean Number of Infiltrating Absolute Cluster of Differentiation 3 (CD3+) T Cells/ μm2
Description: The primary endpoint for this study is the change in the mean number of infiltrating CD3+ T cells/ μm2 in the lung cancer tissue from before and after pembrolizumab +/- SRT by group, based on quantification using immunohistochemistry (IHC) and image analysis by group.
Time Frame: Up to 1 year
Measure: Mean (Full Range); unit: CD3+ T cells/ μm2
Arm/Group | Pembrolizumab + Surgery | Pembrolizumab + Radiation + Surgery
Number analyzed (Participants) | 5 | 4
CD3+ T cells/ μm2 | 2976.00007 [851 to 722704] | 3768.74373 [198 to 879551]

2. Primary Outcome: Percentage of Participants Achieving a Two-fold Increase CD3+ T Cells/μm2
Description: The percentage of participants achieving a two-fold increase from baseline in CD3+ T cells/μm2 will be reported. The goal of achieving a two-fold increase in 40 percent (%) of the evaluable population is a reasonable one, as estimated from a previous study showing greater-than-three-fold increase in 57% of patients when CD3+ T cells/μm2 were measured in prostate cancer tissue treated with a cell- based cancer immunotherapy.
Time Frame: Up to 1 year
Measure: Number; unit: percentage of participants
Arm/Group | Pembrolizumab + Surgery | Pembrolizumab + Radiation + Surgery
Number analyzed (Participants) | 5 | 4
percentage of participants | 40 | 75

3. Secondary Outcome: Percentage of Participants With Treatment-Related Adverse Events (AEs)
Description: Adverse events with an attribution of possible, probable, or definite according to NCI Common Terminology Criteria for Adverse Events (CTCAE) v. 4 including immune-related AEs will be considered treatment related
Time Frame: Up to 1 year
Measure: Number; unit: percentage of participants
Arm/Group | Pembrolizumab + Surgery | Pembrolizumab + Radiation + Surgery
Number analyzed (Participants) | 6 | 6
percentage of participants | 100 | 83.3

4. Secondary Outcome: Percentage of Participants With Grade 3 or Higher Immune-related AEs
Description: Immune-related Adverse events with a Grade of 3 or higher according to NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4 will be reported
Time Frame: Up to 1 year
Measure: Number; unit: percentage of participants
Arm/Group | Pembrolizumab + Surgery | Pembrolizumab + Radiation + Surgery
Number analyzed (Participants) | 6 | 6
percentage of participants | 16.66 | 16.66

5. Secondary Outcome: Median Overall Survival in Months
Description: Overall survival is defined as the time from treatment initiation until death in months with the median and full range reported. Participants lost to follow-up will be censored at the last study visit where survival data was obtained, and those still alive at 12 months will be censored.
Time Frame: Up to 1 year
Population: Censored observations are included in the calculation of the median survival time
Measure: Median (Full Range); unit: months
Arm/Group | Pembrolizumab + Surgery | Pembrolizumab + Radiation + Surgery
Number analyzed (Participants) | 6 | 6
months | 12 [2.13 to 12] | 12 [9.86 to 12]

6. Secondary Outcome: Median Relapse Free Survival
Description: Relapse free survival is defined as the time from treatment initiation until documented disease progression, in months, with the median and full range reported. Participants who have not progressed at the end of 12 months will be censored to the last study visit.
Time Frame: Up to 1 year
Population: Censored observations are included in the calculation of the median survival time
Measure: Median (Full Range); unit: months
Arm/Group | Pembrolizumab + Surgery | Pembrolizumab + Radiation + Surgery
Number analyzed (Participants) | 6 | 6
months | 12 [2.13 to 12] | 12 [9.86 to 12]

7. Secondary Outcome: Percentage of Participants With Distant Metastases
Description: The percentage of participants who demonstrated distant metastases at 12 months will be reported
Time Frame: Up to 1 year
Population: Data not collected
Arm/Group | Pembrolizumab + Surgery | Pembrolizumab + Radiation + Surgery
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Percentage of Participants Determined to Have Unresectable Tumors After Progression
Description: The percentage of participants with demonstrated progression that were determined to have tumor unresectability following the preoperative program will be reported.
Time Frame: Up to 1 year
Measure: Number; unit: percentage of participants
Arm/Group | Pembrolizumab + Surgery | Pembrolizumab + Radiation + Surgery
Number analyzed (Participants) | 6 | 6
percentage of participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 1 year
Arm/Group | Pembrolizumab + Surgery | Pembrolizumab + Radiation + Surgery
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 2/6 | 1/6
Other Adverse Events (participants affected / at risk) | 6/6 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Surgery (N=6) | Pembrolizumab + Radiation + Surgery (N=6)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Surgery (N=6) | Pembrolizumab + Radiation + Surgery (N=6)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hypoxia (Reproductive system and breast disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-29): https://cdn.clinicaltrials.gov/large-docs/71/NCT03217071/Prot_SAP_000.pdf
  • Informed Consent Form (2021-05-12): https://cdn.clinicaltrials.gov/large-docs/71/NCT03217071/ICF_001.pdf